CLINICAL TRIAL: NCT02404155
Title: Biomarker and Safety Study of Clozapine in Patients With Benign Ethnic Neutropenia (BEN)
Acronym: BEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Deanna Kelly, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00063484
Record Dates: First submitted 2015-02-26; First posted 2015-03-31 (Estimated); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clozapine (Experimental)
  Interventions: Drug: Clozapine

INTERVENTIONS:
Drug: Clozapine

SUMMARY:
Clozapine (CLZ) is the most effective antipsychotic for treatment-refractory schizophrenia (SZ). Despite the overwhelming evidence of superior efficacy, CLZ is infrequently prescribed in the US, at a considerably lower rate than the estimated prevalence of treatment-resistant SZ, especially for African-Americans (AA). Recent evidence suggests that low Absolute Neutrophil Counts (ANC), either at baseline or during treatment are a significant barrier to CLZ use in AA patients in the US, where guidelines mandate CLZ discontinuation if ANC drops below 1500 cells/mm3. The investigators group has found that discontinuation of CLZ in AA patients is over twice that in European-American (EA) patients (N~400; 42% vs.19%, P=0.041) and initiation rates are 50% lower. In a Statewide study (N=1875), the investigators reported that discontinuation was more frequently due to neutropenia in the AA sample, though no AA had developed agranulocytosis (8 cases in EA). Benign Ethnic Neutropenia (BEN) in people of African ancestry, including AAs, identifies a group (50% of AA) with low ANCs but no increased risk of agranulocytosis or infection. Low baseline or in-treatment fluctuations requiring CLZ discontinuation under current prescribing guidelines are common in CLZ-treated persons with BEN. In the investigators recent pilot study of N=12 AA patients with BEN, treatment was safely and successfully continued with CLZ despite low baseline ANC (outside current guidelines). Recent evidence implicates a polymorphism in the Duffy Antigen Receptor Chemokine (DARC) gene in the pathophysiology of BEN. In homozygotes (FY-/-) for the DARC null allele, mean within-subject neutrophil counts are reduced, resulting in sporadic ANC <1500 cells/mm3 in 10-15% of people with the allele. In population studies, the FY-/- genotype is found in 0.01% of EAs, 99.3% of sub-Saharan Africans (SSA), and 68% of AAs. Further, a missense DARC mutation has been reported to interact with the DARC FY-/- in determining low WBC in AAs. Normal patterns of week-to-week fluctuation in ANC levels in individuals of African ancestry with BEN and the DARC null genotype are not known, and no published research has examined variation in ANC in African ancestry CLZ-treated SZ patients with BEN and the DARC null genotype (FY-/-). Such data are also lacking on individuals with BEN without the DARC null genotype. Conducting such research will generate genetic marker and safety data that could be used to expand access to CLZ for AA patients who otherwise are eligible to receive this superior treatment option.

ELIGIBILITY:
Inclusion Criteria

* Eligible and recommended for clozapine treatment (e.g. treatment resistant schizophrenia, schizoaffective disorder, bipolar disorder, other psychotic disorder, delusional disorder, hostility, other documented rationale)
* Male or Female
* African Ancestry (African, African-American or African-Caribbean). This population will make up the majority of the study. However, there are cases of BEN in individuals of Middle Eastern, Caucasian, and other ethnicity. The investigators will accept these patients as they may have unknown African ancestry and genotyping will be important.
* Age: 18 to 64 years.
* History of a low absolute neutrophil count (ANC<2500 cells/mm3 in past 24 months)
* Documented ability to sign informed consent. This is a score of ≥10/12 on ESC.
* Effective birth control if of child bearing potential

Exclusion Criteria

* DSM-IV diagnosis of Mental Retardation
* Pregnancy or lactation
* History of myeloproliferative disorder
* Uncontrolled seizure disorder
* History of paralytic ileus
* History of clozapine-induced ANC < 700 mm3
* Systemic Lupus Erythematosus, Multiple Sclerosis, Hashimoto's Thyroiditis, Sjogren's Syndrome, Grave's Disease*
* Medical condition whose pathology or treatment would likely alter the presentation or treatment of schizophrenia or significantly increase the risks associated with the proposed protocol.
* Medical condition affecting patient's ability to mount an immune response
* Current bacterial or viral infection*
* Sickle cell anemia
* Positive for bacteria in urine culture*
* Temperature > 37.5 º Celsius, 99.5 º Fahrenheit*
* Current treated or untreated cancer*
* Documented nutritional deficiencies (such as Beriberi, Pellagra, Rickets, Scurvy, Keshan Disease)*

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 274 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, Pharm.D, BCPP, Principal Investigator — Principal Investigator
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

REFERENCES:
- [Derived] Cavaliere VS, Glassman M, DiPaula BA, Mackowick M, Wehring HJ, Liu F, Chen S, Park J, Love RC, Richardson CM, Vyas G, Kearns AM, Kelly DL. Anti-aggressive effects of clozapine in involuntarily committed black patients with severe mental illness. Schizophr Res. 2022 May;243:163-169. doi: 10.1016/j.schres.2022.03.006. Epub 2022 Mar 28. PMID 35358857
- See also: Maryland Psychiatric Research Center — http://www.mprc.umaryland.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Clozapine: Clozapine
Period: Overall Study
Arm/Group | Clozapine
Started | 274
Completed | 227
Not Completed | 47

BASELINE CHARACTERISTICS:
Arm/Group | Clozapine
Number analyzed (Participants) | 274
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 274
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 137
  Unknown or Not Reported | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 255
  White | 6
  More than one race | 11
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 150
  Nigeria | 124

OUTCOME MEASURES:

1. Primary Outcome: Change in White Blood Cell (WBC) (mm3) and Absolute Neutrophil Counts (ANC) (mm3) in Persons According to Presence of the DARC Null Allele.
Time Frame: 24 week period baseline and endpoint
Population: Genetic information was only able to be collected and analyzed on 249 of t he 274 overall participants.
Measure: Mean (Standard Deviation); unit: cells/mm3
Arm/Group | Clozapine
Number analyzed (Participants) | 249
cells/mm3
  Baseline ANC for CC genotype: number analyzed (Participants) | 199
  Baseline ANC for CC genotype | 2755.1 (1271.5)
  Endpoint ANC for CC genotype: number analyzed (Participants) | 199
  Endpoint ANC for CC genotype | 3079.9 (1563.0)
  Baseline ANC for CT genotype: number analyzed (Participants) | 50
  Baseline ANC for CT genotype | 4360.6 (1779.0)
  Endpoint ANC for CT genotype: number analyzed (Participants) | 50
  Endpoint ANC for CT genotype | 4450.3 (2398.0)
  Baseline WBC for CC genotype: number analyzed (Participants) | 199
  Baseline WBC for CC genotype | 5478.9 (1688.1)
  Endpoint WBC for CC genotype: number analyzed (Participants) | 199
  Endpoint WBC for CC genotype | 5766.1 (1946.4)
  Baseline WBC for CT genotype: number analyzed (Participants) | 50
  Baseline WBC for CT genotype | 7802.0 (2142.0)
  Endpoint WBC for CT genotype: number analyzed (Participants) | 50
  Endpoint WBC for CT genotype | 7702.7 (2607.5)

2. Primary Outcome: Number of Episodes of Agranulocytosis (Count).
Time Frame: 6 months
Measure: Number; unit: Episodes
Arm/Group | Clozapine
Number analyzed (Participants) | 274
Episodes | 1

ADVERSE EVENTS:
Time Frame: For each participants 6 months of enrollment
Arm/Group | Clozapine
All-Cause Mortality (participants affected / at risk) | 0/274
Serious Adverse Events (participants affected / at risk) | 19/274
Other Adverse Events (participants affected / at risk) | 264/274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clozapine (N=274)
Prolapsed Rectum (Gastrointestinal disorders) | 1
Stroke (Musculoskeletal and connective tissue disorders) | 2
Seizure (Nervous system disorders) | 2
Pulmonary Emobolism (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Hospitalization for Clinical Worsening (General disorders) | 3
Diverticulitis (Gastrointestinal disorders) | 1
Severe Neutropenia (Blood and lymphatic system disorders) | 1
Dehydration (General disorders) | 3
Urinary Tract Infection (Infections and infestations) | 1
Atypical Neuroleptic Malignant Syndrome/ Drug Fever (General disorders) | 1
Infection/Cellulitis (Infections and infestations) | 2
Pneumonia (General disorders) | 1
Severe Constipation (Gastrointestinal disorders) | 1
Diffuse Ileus (Gastrointestinal disorders) | 1
Pleural Effusion (General disorders) | 1
Unresponsiveness (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clozapine (N=274)
Abdominal Pain (Gastrointestinal disorders) | 91
Anorexia (General disorders) | 51
Bruising (General disorders) | 12
Constipation (Gastrointestinal disorders) | 88
Diarrhea (Gastrointestinal disorders) | 64
Dizziness (General disorders) | 112
Dry Mouth (General disorders) | 65
Enuresis (Gastrointestinal disorders) | 70
Fever (General disorders) | 35
Headache (General disorders) | 86
Insomnia (General disorders) | 53
Malaise (General disorders) | 144
Mucosal (General disorders) | 22
Nausea (Gastrointestinal disorders) | 77
Rash (General disorders) | 36
Restlessness (Nervous system disorders) | 79
Salivation (Endocrine disorders) | 187
Sedation (General disorders) | 145
Stiffness (Musculoskeletal and connective tissue disorders) | 66
Sore Throat (General disorders) | 49
Tremors (Nervous system disorders) | 73
Urticaria (General disorders) | 59
Vomiting (Gastrointestinal disorders) | 61
Weight loss (Gastrointestinal disorders) | 29
Tinnitus (General disorders) | 37
Abnormal Ejaculation/Erectile Dysfunction (General disorders) | 2
Chest Pain (Cardiac disorders) | 6
Diabetes/Hyperglycemia (Metabolism and nutrition disorders) | 3
Disorientation/Confusion (General disorders) | 2
Edema (General disorders) | 2
Myocarditis (Cardiac disorders) | 1
Myoclonus (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT02404155/Prot_SAP_000.pdf